CLINICAL TRIAL: NCT03220945
Title: A Comprehensive Yoga Program (SKY) as an Adjunct Therapy for Prostate Cancer - A Randomized Pilot Study
Brief Title: Comprehensive Yoga Program (SKY) as Adjunct Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Omer Kucuk, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00084607; NCI-2016-00025 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3059-15 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Control group) (No Intervention): Patients may receive yoga instruction for 1 week after post-test 2.
- Arm II (Yoga group) (Experimental): Patients receive yoga instruction over approximately 3 hours daily for 5 days of week 1 and over 2 hours once a week of weeks 2-13.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Receive yoga instruction
  Other Names: Yoga Therapy
  Arms: Arm II (Yoga group)

SUMMARY:
This randomized pilot trial studies the effect of comprehensive yoga program (SKY) in reducing stress, pain, and fatigue, and improving psychological well-being in patients with prostate cancer. SKY is one of the most widely used breathing techniques derived from yoga. SKY Yoga may improve quality of life in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine any change in pain, fatigue and psychological well-being as a result of SKY in prostate cancer (PCa) patients.

II. Assess changes in some physiological parameters in response to SKY in the same subjects, compare these with those from Part 1, and assess whether these translate into clinical effects.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (Control Group): Patients undergo collection of blood, saliva, and hair samples after signing consent (pre-test 1), within 6-8 weeks after pre-test 1 (post-test 1), and within 2-4 months after post-test 1 (post-test 2). Patients may receive yoga instruction for 1 week after post-test 2.

ARM II (Yoga Group): Patients receive yoga instruction over approximately 3 hours daily for 5 days of week 1 and over 2 hours once a week of weeks 2-13. Patients also undergo collection of blood, saliva, and hair samples within 2 months prior to starting yoga instruction, within weeks 2-3, and within weeks 14-15.

ELIGIBILITY:
Inclusion Criteria:

* Having finished radiotherapy at least two months ago
* Ability to speak and read English and give informed consent
* Have an interest in being part of a study to evaluate yoga-derived exercises and eager to practice some kind of relaxation exercise daily for 3 months

Exclusion Criteria:

* Have a diagnosis of psychiatric illness or other major illness in addition to PCa, such as other cancers, uncontrolled hypertension, lung disease, liver disease or heart disease

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Change in the anxiety and depression, as defined in Hospital Anxiety and Depression Scale (HADS) | 15 weeks after study start
  HADS is a 14-item self-rating scale that measures anxiety and depression. HADS will be compared before and after intervention.
Change in global health-status/QOL scale symptoms as defined in the EORTC Quality-of-life Questionnaire (EORTC QLQ-C30) | 15 weeks after study start
  European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQ-C30) is a cancer-specific 30-item questionnaire incorporating 5-functioning scales, a global health-status/QOL scale and symptoms assessment.
Change in psychological well-being as defined in the Life Orientation Test-Revised (LOT-R) | 15 weeks after study start
  LOT-R is a 10-item self-report scale that measures the expectations about positive outcome in general.
Change in fatigue as defined in 36-item short-form health survey (SF-36) vitality scale | 15 weeks after study start
  SF-36 is a reliable and valid measure of energy/fatigue in the past month.
Change in pain based on brief pain inventory - short form | 15 weeks after study start
  Pain will be assessed with the brief pain inventory - short form (BPI-SF) questionnaire.

SECONDARY OUTCOMES:
Change in antioxidant status: superoxide dismutase | 15 weeks after study start
  Change in the enzyme indicative of antioxidant status, superoxide dismutase, will be assessed.
Change in antioxidant status: glutathione peroxidase | 15 weeks after study start
  Change in the enzyme indicative of antioxidant status, glutathione peroxidase, will be assessed.
Change in serum 8-isoprostane | 15 weeks after study start
  Serum 8-isoprostane level will also be measured as an indicator of oxidative stress.
Change in saliva cortisol | 15 weeks after study start
  Change in saliva cortisol will be compared before and after the intervention to assess the psychophysiological stress.
Change in hair cortisol | 15 weeks after study start
  Change in hair cortisol will be assessed as a measure of psychophysiological stress using a 1-inch strand of hair taken from the back of the head.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03220945/Prot_SAP_001.pdf
  • Informed Consent Form (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03220945/ICF_000.pdf